CLINICAL TRIAL: NCT06295952
Title: Pasireotide Treatment for Patients With Prolactinomas Who Need Treatment Beyond Dopamine Agonist Therapy
Brief Title: A Study of Pasireotide in People With Prolactinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-371
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Prolactin-Producing Pituitary Tumor
Keywords: pasireotide; dopamine agonist; 23-371
MeSH Terms: interventions — pasireotide; 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Intervention Model Description: This is an open label single-center pilot study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pasireotide (Experimental): All patients will initiate open-label treatment with pasireotide LAR on week 1 in the outpatient setting. Pasireotide will be initiated at 40 mg IM one time dose and if tolerated dose will be increased to 60 mg IM every 4 weeks +/-7 days. Administration of pasireotide will align with package inset. Patients must return to the study center every 28 days (+/- 7 days) to receive study medication and for evaluation.
  Interventions: Drug: Pasireotide; Other: SF-36 and HADS

INTERVENTIONS:
Drug: Pasireotide — Pasireotide will be initiated at 40 mg IM one time dose and if tolerated dose will be increased to 60 mg IM every 4 weeks +/-7 days.
Other: SF-36 and HADS — Baseline assessment will be conducted within 30 days of starting treatment, week 12, 24 and week 28.

SUMMARY:
The researchers are doing this study to find out whether pasireotide is an effective treatment for people with prolactinoma who cannot receive dopamine agonist therapy. Another purpose of this study is to find out whether pasireotide is a safe treatment for people with prolactinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Male and female patients with prolactinomas with at least one of the following criteria:

   * Clinical intolerance due to adverse events on DA treatment, preventing continued treatment.
   * Contraindication to DA treatment (e.g., patients requiring dopamine antagonist therapy or other therapy that is contraindicated).
   * Tumor resistance to DA, defined as <50% decrease in longest diameter, or progression in tumor size and/or lack of prolactin normalization with at least 2 mg per week, or maximally tolerated dose, of cabergoline or bromocriptine. Patients with a partial response to DA, including a prolactin reduction but not normalization on treatment, will be included, and will continue DA during the study.
3. Patients are not considered candidates for surgery (e.g., poor surgical candidates, inoperable tumors, patients who refuse surgical treatment, or for whom surgery is deemed not appropriate treatment).
4. For patients with a history of pituitary radiation, the following criteria must be present:

   * At least 6 months must have elapsed from the time of the most recent radiation treatment to the time of enrollment, and
   * Stable or up trending serum prolactin levels and/or evidence of tumor growth since completion of radiation.
5. At least 8 weeks washout of prior first-generation somatostatin receptor ligand therapy (octreotide or lanreotide).
6. Patients on temozolomide will need a washout period of at least 3 weeks.
7. Patients on carboplatin, cisplatin or etoposide will need a washout period of at least 4 weeks.
8. Patients on protein kinase inhibitors (e.g., everolimus, lapatinib) will need a washout period of at least 5 half-lives or 2 weeks, whichever in longer.
9. In general, at least 4 weeks must have elapsed from any other anticancer drug therapy (e.g., bevacizumab).
10. Stable or lower dose of DA (cabergoline or bromocriptine) for at least one month for those patients continuing DA treatment, i.e. DA dose may not be escalated during trial enrollment.
11. Screening laboratory values must meet the following criteria:

    * WBC ≥ 2000/μL
    * Neutrophils ≥ 1500/μL
    * Platelets ≥ 100 x103/μL
    * Hemoglobin > 9.0 g/dL
    * AST/ALT ≤ 3 x ULN
    * Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
    * Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min using the Cockcroft-Gault formula
12. Karnofsky Performance Status (KPS) 70 or above
13. Measurable tumor by RECIST V1.1 criteria, ≥ 10 mm.
14. Women of childbearing potential (WOCBP) must use appropriate methods of contraception while participating in the trial until 30 days after the follow-up period.

    * WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. Women who are not of childbearing potential are not required to use contraception.
    * Women of childbearing potential must have a negative serum or urine pregnancy test upon study entry.
15. Men who are sexually active with women of childbearing potential must use adequate contraception while participating in the trial. Men who are surgically sterile or azoospermia do not require contraception.

Exclusion Criteria:

1. Additional pituitary tumor directed therapy, including temozolomide, everolimus, lapatinib, or cytotoxic chemotherapy
2. Concurrent malignancy except non-melanoma skin cancer
3. Any pituitary surgery within 14 days of enrollment.
4. Patients with poorly controlled diabetes as defined by HBA1c >9% or not optimally treated for diabetes mellitus as judged by the investigator
5. Patients who are not euthyroid as judged by the investigator
6. Patient with liver disease such as cirrhosis, chronic active hepatitis, or chronic persistent hepatitis, or patients with serum ALT and/or AST >3x ULN, or total bilirubin >1.5 x ULN
7. Patients with QTc > 500 ms
8. History of intolerance or resistance to pasireotide
9. Women who are pregnant or breast-feeding
10. Inability to undergo radiographic surveillance
11. Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
biochemical response rate | within 24 weeks of treatment
  response rate as defined by a normal serum prolactin concentration (<18.0 ng/ml for a male and < 29.0 ng/ml for a female

SECONDARY OUTCOMES:
radiographic response | within 24 weeks of treatment
  RECIST criteria, V1.1 (30% decrease in longest tumor diameter)

CONTACTS AND LOCATIONS:
Overall Officials: Eliza Geer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm